CLINICAL TRIAL: NCT03652181
Title: CASH (Cavernous Angiomas With Symptomatic Hemorrhage) Trial Readiness
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Mayo Clinic (Other); Johns Hopkins University (Other); University of California, San Francisco (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Utah (Other); University of New Mexico (Other); Barrow Neurological Institute (Other)
Responsible Party: Sponsor
Other Study IDs: U01NS104157 (NIH); U01NS104157 (NIH)
Record Dates: First submitted 2018-07-18; First posted 2018-08-29 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: CCM; Cavernoma; Cerebral Cavernous Malformation; Cerebral Cavernous Malformations 1; Cerebral Cavernous Malformations 2; Cerebral Cavernous Malformations 3; Cavernous Angioma
Keywords: CCM (Cerebral Cavernous Malformations); Dynamic Contrast Enhanced Quantitative Perfusion (DCEQP); Quantitative Susceptibility Mapping (QSM); Cerebral Cavernous Malformation; Cavernoma; Cavernous Angioma
MeSH Terms: conditions — Hemangioma, Capillary; Hemangioma, Cavernous, Central Nervous System; Cerebral Cavernous Malformations 2; Cerebral Cavernous Malformations 3; Hemangioma, Cavernous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CASH (Cavernous Angiomas with Symptomatic Hemorrhage): The adjudicated definition of CASH (Cavernous Angiomas with Symptomatic Hemorrhage) requires diagnostic evidence of new lesional bleeding or hemorrhagic growth, in association with directly attributable symptoms.

SUMMARY:
Brain Cavernous Angiomas with Symptomatic Hemorrhage (CASH) are rare, but they exact a heavy burden of neurologic disability from recurrent bleeding, for which there is no proven therapy. This trial readiness project aims to address current critical obstacles in identifying cases at multiple sites, characterizing their relevant features, and measuring their outcome. The timing cannot be more opportune, with therapeutic targets already identified, exceptional collaboration among researchers and with the patient community, and several drugs ready to benefit from a track to clinical testing in the next five years.

DETAILED DESCRIPTION:
The Trial Readiness grant mechanism, funded by NINDS, proposes to address knowledge gaps and establish a research network as infrastructure for future research. This project includes an observational cohort study of 181 patients with an operational goal of demonstrating the feasibility of screening, enrollment rates, baseline disease categorization and follow-up of CASH using common data elements at multiple sites, and to assess the following endpoints for 123 participants enrolled at centers prespecified to do prospective follow-up: (1) the rates of recurrent hemorrhage; (2) the reliability of imaging biomarkers including quantitative susceptibility mapping and permeability measures which have been shown to correlate with lesion activity, and (3) change in functional status during prospective follow-up.

ELIGIBILITY:
Inclusion Criteria

1. 18 years of age and older
2. Diagnosed with a brain CA (single or multiple)
3. Had a SH within the past year (with demonstrated new lesional bleeding or hemorrhagic growth on diagnostic studies AND attributable new symptoms)
4. Subject is able to provide informed consent

Exclusion Criteria

1. Spinal CA as source of SH
2. Prior brain irradiation
3. Cases where verification of SH with clinical and imaging review cannot be accomplished
4. Prior or planned treatment of the symptomatic lesion (after neurosurgical consultation)

To be eligible for Aims 2 and 3, CASH cases enrolled in Aim 1 will be further excluded from follow-up and baseline validation (FUBV) for the following reasons:

1. Contraindication for administration of contrast agent or otherwise unwilling or unable to undergo research MRI studies
2. Pregnant or breastfeeding women
3. Homeless or incarcerated persons, or other reason a subject will be unable/unlikely to return for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Brain Cavernous Angiomas with Symptomatic Hemmhorage (CASH) that have occurred within the last year.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam A Awad, MD, Principal Investigator — University of Chicago; Daniel Hanley, MD, Principal Investigator — Johns Hopkins University; Kelly Flemming, MD, Principal Investigator — Mayo Clinic; Helen Kim, MPH, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol has been published in Neurosurgery
Supporting Information: Study Protocol
Time Frame: Protocol paper was published November 2018 in Neurosurgery
Access Criteria: can be accessed through Neurosurgery or Pubmed. Primary study contacts can also provide a copy upon request.

REFERENCES:
- [Derived] Kinkade S, Li H, Hage S, Koskimaki J, Stadnik A, Lee J, Shenkar R, Papaioannou J, Flemming KD, Kim H, Torbey M, Huang J, Carroll TJ, Girard R, Giger ML, Awad IA. Identifying features of prior hemorrhage in cerebral cavernous malformations on quantitative susceptibility maps: a machine learning pilot study. J Neurosurg. 2025 Jul 4;143(6):1567-1574. doi: 10.3171/2025.3.JNS243051. Print 2025 Dec 1. PMID 40614265
- [Derived] Flemming KD, Kim H, Hage S, Mandrekar J, Kinkade S, Girard R, Torbey M, Huang J, Huston J 3rd, Shu Y, Lanzino G, Selwyn R, Hart B, Mabray M, Feghali J, Sair HI, Narvid J, Lupo JM, Lee J, Stadnik A, Alcazar-Felix RJ, Shenkar R, Lane K, McBee N, Treine K, Ostapkovich N, Wang Y, Thompson R, Koenig JI, Carroll T, Hanley D, Awad I. Trial Readiness of Cavernous Malformations With Symptomatic Hemorrhage, Part I: Event Rates and Clinical Outcome. Stroke. 2024 Jan;55(1):22-30. doi: 10.1161/STROKEAHA.123.044068. Epub 2023 Dec 22. PMID 38134268
- [Derived] Hage S, Kinkade S, Girard R, Flemming KD, Kim H, Torbey MT, Huang J, Huston J 3rd, Shu Y, Selwyn RG, Hart BL, Mabray MC, Feghali J, Sair HI, Narvid J, Lupo JM, Lee J, Stadnik A, Alcazar-Felix RJ, Shenkar R, Hobson N, DeBiasse D, Lane K, McBee NA, Treine K, Ostapkovich N, Wang Y, Thompson RE, Koenig JI, Carroll T, Hanley DF Jr, Awad IA. Trial Readiness of Cavernous Malformations With Symptomatic Hemorrhage, Part II: Biomarkers and Trial Modeling. Stroke. 2024 Jan;55(1):31-39. doi: 10.1161/STROKEAHA.123.044083. Epub 2023 Dec 22. PMID 38134265
- [Derived] Hage S, Kinkade S, Girard R, Flemming KD, Kim H, Torbey MT, Huang J, Huston J, Shu Y, Selwyn RG, Hart BL, Mabray MC, Feghali J, Sair HI, Narvid J, Lupo JM, Lee J, Stadnik A, Alcazar R, Shenkar R, Hobson N, DeBiasse D, Lane K, McBee N, Treine K, Ostapkovich N, Wang Y, Thompson RE, Mendoza-Puccini C, Koenig J, Carroll T, Hanley DF, Awad IA. Cavernous Angioma Symptomatic Hemorrhage (CASH) Trial Readiness II: Imaging Biomarkers and Trial Modeling. medRxiv [Preprint]. 2023 Jun 5:2023.06.01.23290854. doi: 10.1101/2023.06.01.23290854. PMID 37333396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 123 participants were enrolled and followed up for 2 years and all results are provided only for these participants.
Period: Overall Study
Arm/Group | CASH (Cavernous Angiomas With Symptomatic Hemorrhage)
Started | 123
Completed Year 1 | 102
Completed Year 2 | 69
Completed | 123
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics will be provided for only those participants who had follow-up.
Arm/Group | CASH (Cavernous Angiomas With Symptomatic Hemorrhage)
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 99
  More than one race | 5
  Unknown or Not Reported | 3
Familial cavernous malformation syndrome [Count of Participants; unit: Participants] — Population: Data were missing for 2 participants
  Participants
    number analyzed (Participants) | 121
    (all) | 48
History of hypertension [Count of Participants; unit: Participants] | 35
History of diabetes [Count of Participants; unit: Participants] | 6
Tobacco use [Count of Participants; unit: Participants] | 11
Obstructive sleep apnea [Count of Participants; unit: Participants] — Population: Data were missing for 12 participants
  Participants
    number analyzed (Participants) | 111
    (all) | 10
Alcohol use [Count of Participants; unit: Participants] | 56
Statin use [Count of Participants; unit: Participants] | 25
Vitamin D supplementation [Count of Participants; unit: Participants] | 88
Propranolol [Count of Participants; unit: Participants] | 7
Birth control [Count of Participants; unit: Participants] — Population: 75 participants were females for whom birth control could be assessed
  Participants
    number analyzed (Participants) | 75
    (all) | 2
Systolic blood pressure, mm Hg [Mean (Standard Deviation); unit: mmHg] — Population: Data were missing for 8 participants
  mmHg
    number analyzed (Participants) | 115
    (all) | 122.7 (14.7)
Diastolic blood pressure, mm Hg [Mean (Standard Deviation); unit: mmHg] — Population: Data were missing for 8 participants
  mmHg
    number analyzed (Participants) | 115
    (all) | 78.3 (10.0)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (5.1)
Qualifying Symptomatic Hemorrhage (SH) location: Brainstem [Count of Participants; unit: Participants]
  Brainstem | 50
  Thalamus | 13
  Lobar | 35
  Cerebellum | 12
  Other | 13

OUTCOME MEASURES:

1. Primary Outcome: Rate of Recurrent Symptomatic Hemorrhage During the Two Year Follow-up Period in Patients With CASH.
Description: Number of new bleeds reported during the two year follow-up period in the cohort with CASH. We will assess the change in the number of new symptomatic hemorrhage from baseline to year 1 and year 1 to year 2 follow-up.
Time Frame: 2 year
Measure: Number; unit: Number of new bleeds
Groups:
- Baseline to Year 1: Change assessed from baseline to Year 1. A total of 102 participants completed year 1 follow-up.
- Year 1 to Year 2: Change assessed from year 1 to year 2
Arm/Group | Baseline to Year 1 | Year 1 to Year 2
Number analyzed (Participants) | 102 | 69
Number of new bleeds | 10 | 11

2. Secondary Outcome: Percent Change in QSM Value (Lesional Iron Content)
Description: Change in QSM value (lesional iron content) will be presented as a mean value across all participants from baseline to year 1 and year 1 to year 2 follow-up MRIs
Time Frame: 2 years of follow-up
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Baseline to Year 1: Change assessed from baseline to Year 1. A total of 102 participants completed year 1 follow-up. Of the 102, 95 had a QSM acquisition of which 93 were usable.
- Year 1 to Year 2: Change assessed from year 1 to year 2. A total of 69 participants completed year 2 follow-up. Of the 69, 59 had a QSM acquisition, of which 56 were usable.
Arm/Group | Baseline to Year 1 | Year 1 to Year 2
Number analyzed (Participants) | 93 | 56
percent change | 16.33 (74.93) | 19.61 (70.96)
Statistical Analysis 1: Comparison: Baseline to Year 1 vs Year 1 to Year 2; Test type: Equivalence — The null hypothesis is that the year 1 change is equivalent to year 2 change in mean QSM; p = 0.033, t-test, 2 sided

3. Secondary Outcome: Percent Change in Contrast-enhanced Quantitative Perfusion (DCEQP) Value (Vascular Permeability)
Description: Change in DCEQP value (vascular permeability) will be presented as a mean value across all participants from baseline to year 1 and year 1 to year 2 follow-up MRIs
Time Frame: 2 years of follow-up
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Baseline to Year 1: Change assessed from baseline to Year 1. A total of 102 participants completed year 1 follow-up. Of the 102, 95 had a DCEQP acquisition of which 85 were usable.
- Year 1 to Year 2: Change assessed from year 1 to year 2. A total of 69 participants completed year 2 follow-up. Of the 69, 59 had a DCEQP acquisition, of which 55 were usable.
Arm/Group | Baseline to Year 1 | Year 1 to Year 2
Number analyzed (Participants) | 85 | 55
percent change | 61.62 (248.8) | 52.45 (206.4)
Statistical Analysis 1: Comparison: Baseline to Year 1 vs Year 1 to Year 2; Test type: Equivalence — The null hypothesis is that the year 1 change is equivalent to year 2 change in mean DCEQP; p = 0.3459, t-test, 2 sided

4. Secondary Outcome: Compare the Number of Patients With MRS 2 or Higher Who Had Prospective Symptomatic Hemorrhage to Those With MRS 2 or Higher Without Prospective Symptomatic Hemorrhage During the 2 Year Follow-up Period.
Description: Compare the number of patients with MRS 2 or higher who had prospective symptomatic hemorrhage to those with MRS 2 or higher without prospective symptomatic hemorrhage from baseline to year 1 and year 1 to year 2 follow-up periods.
  The mRS is a simple global measure of functional disability. Scores range from 0 (no symptoms) to 6 (death). An mRS score of 0 to 1 is considered a minimal clinical disability, and 0 to 2 is independent.
Time Frame: 2 years of follow-up
Population: At year 1, 5 participants with symptomatic hemorrhage were analyzed, and 97 without symptomatic hemorrhage totaling, 102 participants analyzed. At year 2, 7 participants with symptomatic hemorrhage were analyzed, and 62 without symptomatic hemorrhage, totaling 69 participants analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Year 1 to Year 2: Change assessed from year 1 to year 2. A total of 69participants completed year 2 follow-up.
Arm/Group | Baseline to Year 1 | Year 1 to Year 2
Number analyzed (Participants) | 102 | 69
Participants
  Symptomatic hemorrhage: number analyzed (Participants) | 5 | 7
  Symptomatic hemorrhage | 1 | 2
  No symptomatic hemorrhage: number analyzed (Participants) | 97 | 62
  No symptomatic hemorrhage | 27 | 15
Statistical Analysis 1: Comparison: Baseline to Year 1 vs Year 1 to Year 2; Test type: Equivalence — The null hypothesis is that the year 1 change is equivalent to year 2 numbers; p = 1.0, Chi-squared

5. Secondary Outcome: Percentage of Patients With National Institutes of Health Stroke Scale (NIHSS) 0-4, 5-14 and 14+ During the 2 Year Follow-up Period.
Description: Percentage of patients with National Institutes of Health Stroke Scale (NIHSS) 0-4, 5-14 and 14+ from baseline to year 1 and year 1 to year 2 follow-up periods.
  NIHSS values range from 0 to 42, with stroke severity categorized as mild (0 to 4), moderate (5 to 14), severe (15 to 24), and very severe (≥25). 4-point decline in ischemic stroke clinical trials typically measures functional decline.
Time Frame: 2 years of follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Numbers were assessed at baseline . A total of 123 participants were enrolled.
- Year 1: Numbers were assessed at year 1. A total of 98 participants completed year 1 follow-up.
- Year 2: Numbers were assessed at year 2. A total of 61 participants completed year 2 follow-up.
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 98 | 61
Participants
  NIHSS score 0-4 | 117 | 97 | 61
  NIHSS score 5-14 | 5 | 1 | 0
  NIHSS score 14+ | 1 | 0 | 0

6. Secondary Outcome: Median Score of European Quality of Life Visual Analogue Scale (EQ-VAS) During the 2 Year Follow-up Period.
Description: Median score of European Quality of Life Visual Analogue Scale (EQ-VAS) at baseline, year 1, year 2.
  The EQ-VAS is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Time Frame: 2 years of follow-up
Measure: Median (Full Range); unit: score on a scale
Groups:
- Baseline: Median score was assessed at baseline. A total of 119 participants were enrolled.
- Year 1: Median was assessed at Year 1. A total of 102 participants completed year 1 follow-up.
- Year 2: Median was assessed at Year 2. A total of 68 participants completed year 2 follow-up.
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 119 | 102 | 68
score on a scale | 80 [9 to 100] | 80 [30 to 100] | 80 [35 to 100]

7. Secondary Outcome: Proportion of Patients With No Problems, Mild Problems, or Severe Problems in the "Mobility" Domain of European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3 L) During the 2 Year Follow-up Period.
Description: Proportion of patients with no problems, mild problems, or severe problems in the "Mobility" domain of EQ-5D-3 L will be assessed at baseline, year 1, and year 2 follow-up periods.
  EQ-5D-3 L is a generic tool for Patient Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease and includes 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. There are 3 questions per domain where patients respond if they have no problems, mild, or severe problems.
Time Frame: 2 years of follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Proportion assessed at baseline in each category. A total of 123 participants were enrolled
- Year 1: Proportion assessed at year 1 in each category. A total of 102 participants completed year 1 follow-up.
- Year 2: Proportion assessed at year 2 in each category. A total of 68 participants completed year 2 follow-up.
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 68
Participants
  No problems | 83 | 69 | 44
  Mild problems | 40 | 33 | 24
  Severe Problems | 0 | 0 | 0

8. Secondary Outcome: Proportion of Patients With No Problems, Mild Problems, or Severe Problems in the "Self-care" Domain of European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3 L) During the 2 Year Follow-up Period.
Description: Proportion of patients with no problems, mild problems, or severe problems in the "Self-care" domain of EQ-5D-3 L will be assessed at baseline, year 1, and year 2 follow-up periods.
  EQ-5D-3 L is a generic tool for Patient Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease and includes 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. There are 3 questions per domain where patients respond if they have no problems, mild, or severe problems.
Time Frame: 2 years of follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Year 1: Proportion assessed at year 1 in each category. A total of 102 participants were enrolled.
- Year 2: Proportion assessed at year 2 in each category. A total of 68 participants were enrolled.
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 68
Participants
  No problems | 111 | 95 | 63
  Mild problems | 12 | 7 | 5
  Severe problems | 0 | 0 | 0

9. Secondary Outcome: Proportion of Patients With No Problems, Mild Problems, or Severe Problems in the "Usual Activities" Domain of European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3 L) During the 2 Year Follow-up Period.
Description: Proportion of patients with no problems, mild problems, or severe problems in the "Usual activities" domain of EQ-5D-3 L will be assessed at baseline, year 1, and year 2 follow-up periods.
  EQ-5D-3 L is a generic tool for Patient Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease and includes 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. There are 3 questions per domain where patients respond if they have no problems, mild, or severe problems.
Time Frame: 2 years of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 68
Participants
  No problems | 72 | 66 | 50
  Mild problems | 50 | 34 | 17
  Severe problems | 1 | 2 | 1

10. Secondary Outcome: Proportion of Patients With No Problems, Mild Problems, or Severe Problems in the "Pain / Discomfort" Domain of European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3 L) During the 2 Year Follow-up Period.
Description: Proportion of patients with no problems, mild problems, or severe problems in the "Pain / Discomfort" domain of EQ-5D-3 L will be assessed at baseline, year 1, and year 2 follow-up periods.
  EQ-5D-3 L is a generic tool for Patient Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease and includes 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. There are 3 questions per domain where patients respond if they have no problems, mild, or severe problems.
Time Frame: 2 years of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 68
Participants
  No problems | 63 | 63 | 48
  Mild problems | 51 | 36 | 19
  Severe problems | 9 | 3 | 1

11. Secondary Outcome: Proportion of Patients With No Problems, Mild Problems, or Severe Problems in the "Anxiety / Depression" Domain of European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3 L) During the 2 Year Follow-up Period.
Description: Proportion of patients with no problems, mild problems, or severe problems in the "Anxiety / Depression" domain of EQ-5D-3 L will be assessed at baseline, year 1, and year 2 follow-up periods.
  EQ-5D-3 L is a generic tool for Patient Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease and includes 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. There are 3 questions per domain where patients respond if they have no problems, mild, or severe problems.
Time Frame: 2 years of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 68
Participants
  No problems | 72 | 62 | 49
  Mild problems | 46 | 38 | 19
  Severe problems | 5 | 2 | 0

12. Secondary Outcome: Median T-score for "Anxiety" Domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) During the 2 Year Follow-up Period.
Description: Median T-score for "Anxiety" domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) at baseline, year 1 and year 2.
  PROMIS-29 (Version 2.0) is a generic health-related quality of life measure including 7 domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities).12 Each domain contains questions ranked using a 5-point Likert scale. PROMIS-29 domain scores are converted to T scores and have been standardized to a reference population (mean, 50; SD, 10). Clinically meaningful change is considered to be at least half the SD (5 points). Higher T-score indicates better outcome.
Time Frame: 2 years of follow-up
Measure: Median (Full Range); unit: T-score
Groups:
- Baseline: Median T score was assessed at baseline. A total of 123 participants were enrolled.
- Year 1: Median T score was assessed at Year 1. A total of 102 participants completed year 1 follow-up.
- Year 2: Median T score was assessed at Year 2. A total of 67 participants completed year 2 follow-up.
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 67
T-score | 53.7 [40.3 to 75.4] | 51.2 [40.3 to 69.3] | 51.2 [40.3 to 71.2]

13. Secondary Outcome: Median T-score for "Depression" Domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) During the 2 Year Follow-up Period.
Description: Median T-score for "Depression" domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) at baseline, year 1, and year 2.
  PROMIS-29 (Version 2.0) is a generic health-related quality of life measure including 7 domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities).12 Each domain contains questions ranked using a 5-point Likert scale. PROMIS-29 domain scores are converted to T scores and have been standardized to a reference population (mean, 50; SD, 10). Clinically meaningful change is considered to be at least half the SD (5 points). Higher T-score indicates better outcome.
Time Frame: 2 years of follow-up
Measure: Median (Full Range); unit: T-score
Groups:
- Year 2: Median T score was assessed at Year 2. A total of 67 participants completed year 1 follow-up.
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 67
T-score | 41.0 [41.0 to 71.2] | 41.0 [41.0 to 63.9] | 41.0 [41.0 to 65.7]

14. Secondary Outcome: Median T-score for "Fatigue" Domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) During the 2 Year Follow-up Period.
Description: Median T-score for "Fatigue" domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) at baseline, year 1, and year 2.
  PROMIS-29 (Version 2.0) is a generic health-related quality of life measure including 7 domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities).12 Each domain contains questions ranked using a 5-point Likert scale. PROMIS-29 domain scores are converted to T scores and have been standardized to a reference population (mean, 50; SD, 10). Clinically meaningful change is considered to be at least half the SD (5 points). Higher T-score indicates better outcome.
Time Frame: 2 years of follow-up
Measure: Median (Full Range); unit: T-score
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 67
T-score | 48.6 [33.7 to 75.8] | 48.6 [33.7 to 75.8] | 46.0 [33.7 to 75.8]

15. Secondary Outcome: Median T-score for "Pain" Domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) During the 2 Year Follow-up Period.
Description: Median T-score for "Pain" domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) at baseline, year 1 and year 2.
  PROMIS-29 (Version 2.0) is a generic health-related quality of life measure including 7 domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities).12 Each domain contains questions ranked using a 5-point Likert scale. PROMIS-29 domain scores are converted to T scores and have been standardized to a reference population (mean, 50; SD, 10). Clinically meaningful change is considered to be at least half the SD (5 points). Higher T-score indicates better outcome.
Time Frame: 2 years of follow-up
Measure: Median (Full Range); unit: T-score
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 67
T-score | 49.6 [41.6 to 75.6] | 49.6 [41.6 to 75.6] | 41.6 [41.6 to 71.6]

16. Secondary Outcome: Median T-score for "Sleep Disturbance" Domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) During the 2 Year Follow-up Period.
Description: Median T-score for "Sleep Disturbance" domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) at baseline, year 1 and year 2.
  PROMIS-29 (Version 2.0) is a generic health-related quality of life measure including 7 domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities).12 Each domain contains questions ranked using a 5-point Likert scale. PROMIS-29 domain scores are converted to T scores and have been standardized to a reference population (mean, 50; SD, 10). Clinically meaningful change is considered to be at least half the SD (5 points). Higher T-score indicates better outcome.
Time Frame: 2 years of follow-up
Measure: Median (Full Range); unit: T-score
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 67
T-score | 50.5 [43.8 to 61.7] | 50.5 [43.8 to 63.8] | 50.5 [43.8 to 63.8]

17. Secondary Outcome: Median T-score for "Social" Domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) During the 2 Year Follow-up Period.
Description: Median T-score for "Social" domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) at baseline, year 1 and year 2.
  PROMIS-29 (Version 2.0) is a generic health-related quality of life measure including 7 domains (anxiety, depression, fatigue, pain interference, sleep disturbance, and ability to participate in social roles and activities, and physical function).12 Each domain contains questions ranked using a 5-point Likert scale. PROMIS-29 domain scores are converted to T scores and have been standardized to a reference population (mean, 50; SD, 10). Clinically meaningful change is considered to be at least half the SD (5 points). Higher T-score indicates better outcome.
Time Frame: 2 years of follow-up
Measure: Median (Full Range); unit: T-score
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 67
T-score | 51.9 [27.5 to 64.2] | 51.9 [27.5 to 64.2] | 64.2 [34.0 to 64.2]

18. Secondary Outcome: Median T-score for "Physical Function" Domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) During the 2 Year Follow-up Period.
Description: Median T-score for "Physical Function" domain of Patient-Reported Outcome Measurement Information System (PROMIS-29) at baseline, year 1 and year 2.
  PROMIS-29 (Version 2.0) is a generic health-related quality of life measure including 7 domains (anxiety, depression, fatigue, pain interference, sleep disturbance, and ability to participate in social roles and activities, and physical function).12 Each domain contains questions ranked using a 5-point Likert scale. PROMIS-29 domain scores are converted to T scores and have been standardized to a reference population (mean, 50; SD, 10). Clinically meaningful change is considered to be at least half the SD (5 points). Higher T-score indicates better outcome.
Time Frame: 2 years of follow-up
Measure: Median (Full Range); unit: T-score
Arm/Group | Baseline | Year 1 | Year 2
Number analyzed (Participants) | 123 | 102 | 67
T-score | 56.9 [22.9 to 56.9] | 56.9 [26.9 to 56.9] | 56.9 [30.7 to 56.9]

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed for this study since it is an observational study for trial readiness.
Description: Adverse events were not assessed for this study since it is an observational study for trial readiness.
Arm/Group | CASH (Cavernous Angiomas With Symptomatic Hemorrhage)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT03652181/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03652181/ICF_001.pdf